CLINICAL TRIAL: NCT04862065
Title: Alinity s Anti-HCV II - Clinical Evaluation Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Transfusion Medicine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: T3M3-02-19H04-01
Record Dates: First submitted 2021-04-23; First posted 2021-04-27 (Actual); Results first posted 2022-09-16 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-09

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Evaluation of assay performance characteristics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Screening (Other): Alinity s Anti-HCV and Alinity s Anti-HCV II. A follow-up visit may be needed if investigational Alinity s Anti-HCV II result is discordant after supplemental testing.
  Interventions: Device: Alinity s Anti-HCV II

INTERVENTIONS:
Device: Alinity s Anti-HCV II — For all donor specimens with investigational Alinity s Anti-HCV II results that are discordant with final status after supplemental testing, an attempt will be made to obtain a follow-up whole blood specimen approximately 4 to 6 weeks after initial donation for further analysis.

SUMMARY:
The objective of this study is to demonstrate the performance and intended use of the Alinity s Anti-HCV II investigational assay in a donor screening environment using clinical samples to evaluate assay performance. The Alinity s Anti-HCV II assay performance will be evaluated utilizing the Food and Drug Administration (FDA) licensed Alinity s Anti-HCV assay as the comparator method. The data will be used to support regulatory submissions and/or publications.

DETAILED DESCRIPTION:
This study evaluates the Alinity s Anti-HCV II investigational assay using the Alinity s System.

The Alinity s Anti-HCV II assay is a chemiluminescent microparticle immunoassay (CMIA) used for the qualitative detection of antibodies to hepatitis C virus (HCV) in human serum and plasma specimens on the Alinity s System. The Alinity s Anti-HCV II assay is intended to screen individual human donors, including volunteer donors of whole blood and blood components, and other living donors for the presence of anti-HCV.

The performance of the Alinity s Anti-HCV II assay will be evaluated by performing specificity, and sensitivity testing of the Alinity s Anti-HCV II assay.

To evaluate specificity, approximately 15,000 random unique donor specimens will be collected.

To evaluate sensitivity, Abbott will provide a minimum of 400 frozen samples from U.S. individuals characterized as HCV positive and a minimum of 400 frozen specimens from U.S. individuals at increased risk for HCV infection.

ELIGIBILITY:
Inclusion Criteria:

* Serum or ethylenediaminetetraacetic acid (EDTA) plasma from a blood donor or a plasma from a plasmapheresis donor.

Exclusion Criteria:

* Previous participation in this study. Each subject must be represented only once in the study.

Note: Frozen samples (sensitivity) provided by Abbott (403 specimens characterized as positive for HCV and 404 specimens with Increased risk of HCV infection) have no specific inclusion/exclusion criteria that the clinical sites need to verify prior to testing. Inclusion and exclusion criteria only apply to specificity specimens.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16388 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theresa A Nester, MD, Principal Investigator — Bloodworks Northwest; Thomas S Jones, Ph.D., Principal Investigator — QualTex Laboratories; Toby L Simon, M.D., Principal Investigator — CSL Plasma Inc.; Jed Gorlin, M.D., Principal Investigator — Innovative Blood Resources
Locations (4):
- United States (4):
  - Innovative Blood Resources, Saint Paul, Minnesota
  - CSL Plasma Inc., Knoxville, Tennessee
  - QualTex Laboratories, San Antonio, Texas
  - Bloodworks Northwest, Renton, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Alinity s Anti-HCV II: 16,388
Groups:
- Specificity: US blood and/or plasmapheresis donor specimens collected as part of routine blood and/or plasma donation were tested with the investigational Alinity s Anti-HCV II assay.
- Sensitivity: Specimens characterized as positive for hepatitis C virus (HCV) obtained from specimen vendors were tested by the investigational Alinity s Anti-HCV II assay.
- Increased Risk Population: Specimens with Increased Risk of Infection for hepatitis C virus (HCV) obtained from specimen vendors were tested with investigational Alinity s Anti-HCV II assay.
Period: Screening
Arm/Group | Specificity | Sensitivity | Increased Risk Population
Started | 15581 | 403 | 404
Completed | 15526 | 403 | 404
Not Completed | 55 | 0 | 0
Not completed — Protocol Violation | 54 | 0 | 0
Not completed — Insufficient Sample | 1 | 0 | 0
Period: Follow-Up
Arm/Group | Specificity | Sensitivity | Increased Risk Population
Started | 6 | 0 | 0
Completed | 3 | 0 | 0
Not Completed | 3 | 0 | 0
Not completed — Lost to Follow-up | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Units Other Than Participants: Specimens
Groups:
- Sensitivity: Specimens characterized as positive obtained from specimen vendors were tested by the investigational Alinity s Anti-HCV II assay.
- Increased Risk Population: Specimens with Increased Risk of Infection obtained from specimen vendors were tested with investigational Alinity s Anti-HCV II assay.
- Total: Total of all reporting groups
Arm/Group | Specificity | Sensitivity | Increased Risk Population | Total
Number analyzed (Participants) | 15,581 | 403 | 404 | 16388
Number analyzed (Specimens) | 15581 | 403 | 404 | 16388
Age, Customized [Count of Units; unit: Specimens]
  ≥18 Years old | 15,580 | 397 | 404 | 16381
  17 Years old | 1 | 2 | 0 | 3
  16 Years old | 0 | 2 | 0 | 2
  6 Years old | 0 | 1 | 0 | 1
  3 Years old | 0 | 1 | 0 | 1
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 0 | 271 | 247 | 518
  Female | 0 | 132 | 157 | 289
  Unknown | 15,581 | 0 | 0 | 15581
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 38 | 35 | 73
  Not Hispanic or Latino | 0 | 90 | 369 | 459
  Unknown or Not Reported | 15,581 | 275 | 0 | 15856
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Hispanic or Latino counted under Ethnicity section
  Participants
    number analyzed (Participants) | 15,581 | 365 | 369 | 16315
    American Indian or Alaska Native | 0 | 2 | 1 | 3
    Asian | 0 | 2 | 2 | 4
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 0 | 43 | 262 | 305
    White | 0 | 38 | 88 | 126
    More than one race | 0 | 5 | 14 | 19
    Unknown or Not Reported | 15,581 | 275 | 2 | 15858
Region of Enrollment [Number; unit: participants]
  United States | 15,581 | 403 | 404 | 16388

OUTCOME MEASURES:

1. Primary Outcome: Assay Specificity Results for Participants (Specimens) Tested With Alinity s Anti-HCV II Assay.
Description: A total of 15,526 serum and plasma specimens from whole blood donors as well as plasmapheresis specimens were tested with the investigational Alinity s Anti-HCV II assay. Repeatedly reactive specimens were tested further with supplemental assays, if required, to determine final status.
  Anti-HCV II Repeatedly Reactive, Final Status Indeterminate = B
  Anti-HCV II Repeatedly Reactive, Final Status Negative = C
  Anti-HCV II Nonreactive, Final Status Negative = F
  Specificity is calculated as the proportion of nonreactive specimens from specimens with negative status: F / (C+F) × 100%
  Specificity can be also calculated as the proportion of nonreactive specimens with negative status from specimens with negative status and repeatedly reactive specimens with indeterminate status: F / (C + B + F) × 100%
Time Frame: Each participant (specimen) was tested on the Alinity s Anti-HCV II assay in 1 day.
Population: 15,526 serum and plasma specimens from whole blood donors as well as plasmapheresis specimens were tested with Alinity s Anti-HCV II assay.
Measure: Count of Units; unit: Specimen
Units Other Than Participants: Specimen
Arm/Group | Specificity
Number analyzed (Participants) | 15,526
Number analyzed (Specimen) | 15526
Specimen
  Alinity s Anti-HCV II Nonreactive, Final Status Negative | 15,506
  Alinity s Anti-HCV II Repeatedly Reactive, Final Status Negative | 6
  Alinity s Anti-HCV II Repeatedly Reactive, Final Status Positive | 14
Statistical Analysis 1: Comparison: Specificity; Test type: Superiority; Binomial Distribution; Specificity sample size is a minimum of 15,000 donors; Clinical Specificity (%) = 99.96, 95% CI 2-sided [99.92 to 99.99]

2. Primary Outcome: Assay Sensitivity Results for Participants (Specimens) Characterized as Positive Tested With Alinity s Anti-HCV II Assay.
Description: A total of 403 specimens characterized as positive for HCV were obtained from specimen vendors and tested with the investigational Alinity s Anti-HCV II assay.
  Anti-HCV II Repeatedly Reactive, Final Status Positive = A
  Anti-HCV II Nonreactive, Final Status Positive = D
  Anti-HCV II Nonreactive, Final Status Indeterminate = E
  Sensitivity is calculated as the proportion of repeatedly reactive specimens from specimens with positive final status: A / (A+D) × 100%
  Sensitivity can also be calculated as the proportion of repeatedly reactive specimens with positive status from specimens with positive status and nonreactive specimens with indeterminate status: A / (A + D + E) × 100%
Time Frame: Each participant (specimen) was tested on the Alinity s Anti-HCV II assay in 1 day.
Population: 403 specimens characterized as positive for Anti-HCV, 3 of which were classified as Acute HCV positive, were tested with Alinity s Anti-HCV II assay.
Measure: Count of Units; unit: Specimen
Units Other Than Participants: Specimen
Groups:
- Sensitivity: Specimens characterized as positive obtained from specimen vendors were tested with the investigational Alinity s Anti-HCV II assay.
Arm/Group | Sensitivity
Number analyzed (Participants) | 403
Number analyzed (Specimen) | 403
Specimen
  Alinity s Anti-HCV II Nonreactive | 0
  Alinity s Anti-HCV II Repeatedly Reactive | 403
Statistical Analysis 1: Comparison: Sensitivity; Test type: Other — 95% Confidence Interval provided; Sensitivity; Point Estimate = 100.00, 95% CI 2-sided [99.09 to 100.00]

3. Secondary Outcome: Assay Sensitivity Results for Participants (Specimens) With Increased Risk for HCV Tested With Alinity s Anti-HCV II Assay.
Description: 404 specimens from subjects at increased risk for HCV infection were obtained from specimen vendors and tested with investigational Alinity s Anti-HCV II assay. Repeatedly reactive specimens were tested further with supplemental assays, if required, to determine final status.
  Anti-HCV II Repeatedly Reactive, Final Status Positive = A
  Anti-HCV II Nonreactive, Final Status Positive = D
  Anti-HCV II Nonreactive, Final Status Indeterminate = E
  Sensitivity is calculated as the proportion of repeatedly reactive specimens from specimens with positive final status: A / (A+D) × 100%
  Sensitivity can also be calculated as the proportion of repeatedly reactive specimens with positive status from specimens with positive status and nonreactive specimens with indeterminate status: A / (A + D + E) × 100%
Time Frame: Each participant (specimen) was tested on the Alinity s Anti-HCV II assay in 1 day.
Population: A total of 404 specimens from subjects known to be at increased risk for HCV infection were obtained from specimen vendors and tested with investigational Alinity s Anti-HCV II assay.
Measure: Count of Units; unit: Specimen
Units Other Than Participants: Specimen
Arm/Group | Increased Risk Population
Number analyzed (Participants) | 404
Number analyzed (Specimen) | 404
Specimen
  Alinity s Anti-HCV II Nonreactive, Final Status Negative | 324
  Alinity s Anti-HCV II Nonreactive, Final Status Positive | 0
  Alinity s Anti-HCV II Nonreactive, Final Status Indeterminate | 0
  Alinity s Anti-HCV II Reactive, Final Status Positive | 70
  Alinity s Anti-HCV II Reactive, Final Status Negative | 10
  Alinity s Anti-HCV II Reactive, Final Status Indeterminate | 0
Statistical Analysis 1: Comparison: Increased Risk Population; Sensitivity; Test type: Other — 95% Confidence Interval provided; Sensitivity; Point Estimate = 100.00, 95% CI 2-sided [94.87 to 100.00]

ADVERSE EVENTS:
Time Frame: Subject adverse events related to blood collection during the 4-6 weeks of donor follow-up specimen collection.
Description: Adverse Events (AE) had to be reported for donors who returned to provide follow-up sample specifically collected for the study.
  Specificity samples were leftover deidentified specimens from routine blood and plasmapheresis donations, not specifically collected for the study. AEs could not be reported for this population.
  Frozen samples provided by Abbott (HCV positive and at increased risk of HCV infection) were obtained from specimen vendors. AEs could not be reported for these populations.
Groups:
- Alinity s Anti-HCV II Follow-Up Specimen Collection: For all donor specimens with investigational Alinity s results that are discordant with final status after supplemental testing, an attempt was made to obtain a follow-up whole blood specimen approximately 4 to 6 weeks after initial donation for further analysis.
  6 donors were eligible for follow-up collection for Alinity s Anti-HCV II study. 3 out of 6 were able to provide follow-up specimen.
Arm/Group | Alinity s Anti-HCV II Follow-Up Specimen Collection
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI must provide a copy of any proposed publication/presentation at least 60 days prior to submission for sponsor's review/approval. The PI must incorporate changes as the sponsor requires in order to protect the sponsor's proprietary rights and interests. The sponsor may require the PI to include acknowledgement of the sponsor's role in the study. The PI may be requested to delay publication/presentation an extra 60 days to enable sponsor to secure patent or other proprietary protection.

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2020-11-16): https://cdn.clinicaltrials.gov/large-docs/65/NCT04862065/Prot_SAP_000.pdf
  • Informed Consent Form: Information Sheet (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/65/NCT04862065/ICF_001.pdf
  • Informed Consent Form: Follow-Up Consent (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/65/NCT04862065/ICF_002.pdf